CLINICAL TRIAL: NCT05413447
Title: Assessment of Digital Consultations on Clinical Impact and Efficiency Using a RCT (ADMINISTER) Trial
Brief Title: Assessment of Digital Consultations on Clinical Impact and Efficiency
Acronym: ADMINISTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Mark Schuuring, Principle investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123456567
Record Dates: First submitted 2022-05-30; First posted 2022-06-10 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
Keywords: Digital consultations, GDMT optimization, HFrEF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Masking the clinicians of the control group assignment is done to optimally capture local practice. Masking of the intervention group is not feasable as patients and healthcare workers will know whether they are receiving normal care or digital care. Outcome measures are determined beforehand.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving digital consultations (Experimental): The intervention group receive multifaceted digital consults including 1) digital data sharing (e.g. exchange of pharmacotherapy use, home measured vital signs, etc), 2) patient education via an eLearning, and 3) digital guideline recommendations to treating physicians. The consultations are performed remotely unless there is an indication to perform the consult physically.
  Interventions: Combination Product: Digital consult
- Standard care (No Intervention): If the patient is drawn into the control group the patient will receive standard care. Clinicians are free to use all standard modes of communication, and are not specifically encouraged to use remote types of communication. The clinicians are not informed about the assignment of a patient to the control group to optimally capture remote practice.

INTERVENTIONS:
Combination Product: Digital consult — Consultations will be prepared digitally using the Mychart patient portal, an elearning and questionnaires. The consultation takes place via Teams.
  Arms: Patients receiving digital consultations

SUMMARY:
Healthcare workers have a high workload as compared to other sectors and this burden is projected to increase due to an aging society. It is and will in the future be challenging to deliver optimal HF care because of personnel shortages, the high costs of healthcare, intensive GDMT uptitration schedules, and an epidemic rise in HF patients.This study aims to evaluate the impact of digital consultations (DC) on efficiency and clinical impact in heart failure (HF) patients.

A randomized controlled trial on multifaceted digital consults including 1) digital data sharing (e.g. exchange of pharmacotherapy use, home measured vital signs, etc), 2) patient education via an eLearning, and 3) digital guideline recommendations to treating physicians. Included patients will be randomly (1:1) assigned to the intervention group or standard care.

The ADMINISTER trial is expected to offer the first robust randomized controlled multicenter data of GDMT prescription rates, time till full GDMT optimization, time spent on healthcare, patient satisfaction and quality of life of digital consults in GDMT optimization.

DETAILED DESCRIPTION:
Introduction: Many heart failure (HF) patients do not receive optimal guideline-directed medical therapy (GDMT) despite clear benefit on morbidity and mortality outcomes. Digital consultations (DC) have the potential to improve efficiency on GDMT optimization to serve the growing HF population. Hence, the investigator initiated ADMINISTER trial was designed as a pragmatic multicenter randomized controlled trial to evaluate efficacy and safety of DC in patients on HF treatment.

Methods: Patients (n = 150) diagnosed with HF with a reduced ejection fraction (HFrEF) will be randomized to DC or standard care (1:1). The intervention group receive multifaceted digital consults including 1) digital data sharing (e.g. exchange of pharmacotherapy use, home measured vital signs, etc), 2) patient education via an eLearning, and 3) digital guideline recommendations to treating physicians. The consultations are performed remotely unless there is an indication to perform the consult physically. The primary outcome is the GDMT prescription rate score, secondary outcomes include time till full GDMT optimization, patient and clinician satisfaction, time spent on healthcare, and Kansas City Cardiomyopathy questionnaire. Results will be reported in accordance to the CONSORT statement.

Conclusion: The ADMINISTER trial will offer the first randomized controlled data on GDMT prescription rates, time till full GDMT optimization, time spent on healthcare, quality of life, and patient and clinician satisfaction of the multifaceted patient and clinician targeted DC for GDMT optimization.

ELIGIBILITY:
Inclusion Criteria:

* HFrEF

Exclusion Criteria:

* Patients not in possession of any attributes to perform the consults digitally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Prescription rate of ACE/ARNI according to the guidelines | 12 weeks after baseline
  The treatment with ACE/ARNI in accordance to the guideline is measured at baseline and within 4 weeks after the consult. The received dose is divided by the target dose per timepoint. The score will range between a maximum of 1 (corresponding with a treatment according to the guidelines) and a minimum of 0 (corresponding with not administering the medicine). Significant differences between the two groups are determined at both timepoints.
Prescription rate of betablockers according to the guidelines | 12 weeks after baseline
  The treatment with betablockers in accordance to the guideline is measured at baseline and within 4 weeks after the consult. The received dose is divided by the target dose per timepoint. The score will range between a maximum of 1 (corresponding with a treatment according to the guidelines) and a minimum of 0 (corresponding with not administering the medicine). Significant differences between the two groups are determined at both timepoints.
Prescription rate of MRA according to the guidelines | 12 weeks after baseline
  The treatment with MRA in accordance to the guideline is measured at baseline and within 4 weeks after the consult. The received dose is divided by the target dose per timepoint. The score will range between a maximum of 1 (corresponding with a treatment according to the guidelines) and a minimum of 0 (corresponding with not administering the medicine). Significant differences between the two groups are determined at both timepoints.
Prescription rate of SGLT2i according to the guidelines | 12 weeks after baseline
  The treatment with SGLT2i in accordance to the guideline is measured at baseline and within 4 weeks after the consult. The received dose is divided by the target dose per timepoint. The score will range between a maximum of 1 (corresponding with a treatment according to the guidelines) and a minimum of 0 (corresponding with not administering the medicine). Significant differences between the two groups are determined at both timepoints.
Prescription rate of periodic screening of iron insufficiency | 12 weeks after baseline
  It is checked whether periodic (once a year) screening of iron deficiency is performed. And if the patient had iron insufficiency; it is checked whether the patient is receiving intravenous iron administration. Iron insufficiency is defined as ferritin <100 ng/ml or ferritin < 300 ng/ml with transferrin saturation (TSAT) < 20%. For patients with periodic screening for iron deficiency and if appropriate supplementation, a score of 1 was assigned. Other patients will receive a score of 0. Significant differences between groups will be assessed at both timepoints.

SECONDARY OUTCOMES:
Patient satisfaction | At baseline and 12 weeks after the baseline recording
  Patient satisfaction measured with the Net Promotor Score. This is a score in which the patient is asked to give a value between 1 and 10 indicating the likelihood that he/she will recommend the care given at the AUMC to other patients (1 equals unlikely and 10 likely).
Difference in summary score of Kansas city cardiomyopathy questionnaire | At baseline and 12 weeks after the baseline recording
  Worsening of experienced HF, assessed with the "Kansas city cardiomyopathy questionnaire". This will lead to a summary score indicating the severity of the experienced heart failure. This score will range from 0 indicating a bad outcome of the questionnaire to 100 indicating a good outcome.
Time spend on healthcare | 12 weeks after baseline
  The amount of time the patient spends on healthcare.
Amount of hospitalizations per patient | Hospitalization are recorded from baseline until 12 weeks after baseline
  Amount of hospitalizations is recorded for each patient and group differences between the treatment and control group are determined
Healthcare satisfaction | 12 weeks after baseline
  Clinicians will be asked to rate their satisfaction using the Net Promotor Score. This is a score in which the clinician is asked to give a value between 1 and 10 indicating the likelihood that he/she will recommend the remote care with digital consultations to other collegues (1 equals unlikely and 10 likely).

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Cardiology Centers of the Netherlands, Amsterdam, North Holland
  - Amsterdam UMC, location VUmc, Amsterdam
  - Red Cross Hospital, Beverwijk
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Man JP, Koole MAC, Meregalli PG, Handoko ML, Stienen S, de Lange FJ, Winter MM, Schijven MP, Kok WEM, Kuipers DI, van der Harst P, Asselbergs FW, Zwinderman AH, Dijkgraaf MGW, Chamuleau SAJ, Schuuring MJ. Digital consults in heart failure care: a randomized controlled trial. Nat Med. 2024 Oct;30(10):2907-2913. doi: 10.1038/s41591-024-03238-6. Epub 2024 Aug 31. PMID 39217271